CLINICAL TRIAL: NCT05201053
Title: Coagulation Disturbances and Thrombosis in Acute Pancreatitis (Koagulopati Och Trombos Vid Akut Pankreatit-APK Studien)
Brief Title: Acute Pancreatitis and Coagulation Study
Acronym: APK
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/490
Record Dates: First submitted 2022-01-04; First posted 2022-01-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Pancreatitis
Keywords: Acute Pancreatitis; biomarkers; severity prediction
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — Serum and plasma. For some patients alveolar fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild acute pancreatitis: Groups are defined by the Revised Atlanta classification. Anticipated 60% mild, 30% moderate and 10% severe patients
  Interventions: Diagnostic Test: Exploratory for different markers
- moderately severe acute pancreatitis: Groups are defined by the Revised Atlanta classification. Anticipated 60% mild, 30% moderate and 10% severe patients
  Interventions: Diagnostic Test: Exploratory for different markers
- severe acute pancreatitis: Groups are defined by the Revised Atlanta classification. Anticipated 60% mild, 30% moderate and 10% severe patients
  Interventions: Diagnostic Test: Exploratory for different markers

INTERVENTIONS:
Diagnostic Test: Exploratory for different markers — Test biomarkers for development of mild, moderate or severe disease

SUMMARY:
The study aims to investigate pathophysiological changes in coagulation in relation to inflammation in patients with acute pancreatitis. Serum and plasma is sampled repeated days from admission. Analysis will be done after recruitment. Specific biomarkers accuracy for prediction of moderate and severer acute pancreatitis will be calculated.

DETAILED DESCRIPTION:
Inclusion criteria:

Patients with acute pancreatitis admitted to Skåne University Hospital in Malmö

Acute pancreatitis is defined as minimum 2 out of following: amylase levels >3 times upper reference limit, clinical signs of acute pancreatitis, imaging findings of acute pancreatitis)

Exclusion criteria:

<18 years of age

>72 hours from onset of symptom until first sampling

Patients with immunosuppression or autoimmune diseases are excluded from som parts of the study.

Methods: Serum and plasma is sampled repeatedly during the hospital admission. Pre defined protocols are used for data collections of relevant clinical information.

Specific aspects of inflammation, thrombin generation, platelet function and Microparticles will be analysed in serum or plasma during the first consecutive days of acute pancreatitis.

Biomarkers for severe disease as well as correlation between inflammation and coagulopathy will be investigated.

ELIGIBILITY:
Inclusion Criteria: Acute Pancreatitis, accept informed consent -

Exclusion Criteria: More than 72h from onset of symptoms until first sample, patient already included once

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with Acute Pancreatitis at Skåne University Hospital in Malmö
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Severe acute pancreatitis | 14 days
  According to Revised Atlanta which is a consensus document where organ failure (defined by modified Marshall score) less than 48hours or signs of local complications on CT scan defines severity. This is not a scale but a generally used definition according to the paper: Banks PA, et al. Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus. Gut.
  2013;62(1):102-11.

SECONDARY OUTCOMES:
Moderately Severe Acute Pancreatitis | 14 days
  According to Revised Atlanta which is a consensus document where organ failure (defined by modified Marshall score) less than 48hours or signs of local complications on CT scan defines severity. This is not a scale but a generally used definition according to the paper: Banks PA, et al. Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus. Gut.
  2013;62(1):102-11.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Regnér, MD, PhD, Principal Investigator — Region Skåne and Lund University
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After publications. Upon request from other researchers or publishers with scientific interest and in accordance with GDPR regulations
Supporting Information: Study Protocol, SAP
Time Frame: During 2023
Access Criteria: Upon request from other researchers or publishers with scientific interest and in accordance with GDPR regulations